CLINICAL TRIAL: NCT04054869
Title: Bio-mechanical Reasoning and Lateral Specificity of Upper Cervical Joint Mobilization to Improve Cervical Rotation, Improve Function and Reduce Pain.... Does it Matter?
Brief Title: Bio-mechanical Reasoning and Lateral Specificity of Upper Cervical Joint Mobilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrews University (Other)
Responsible Party: Principal Investigator, Michael J Williams, Physical Therapist, Andrews University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 19-089
Record Dates: First submitted 2019-08-04; First posted 2019-08-13 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Neck Pain
Keywords: neck stiffness; manual therapy; joint mobilization
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: each participant receives both treatments in randomized order
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and the outcomes assessor will be masked (blinded) as to the order in which each participant receives the interventions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-mechanically correct manual therapy (received first) arm (Experimental): Participants will be randomized to receive manual therapy directed at the cervical spine atlanto-axial joints in the bio-mechanically correct direction followed by instruction in a home program to maintain this motion. Outcome measures will be assessed. Participants will return in 2-3 days and receive the opposite treatment and home program followed by outcomes assessment. Participants will return again in 2-3 days, outcomes will be assessed and the study will conclude. Participants will then be given the option to continue in formalized physical therapy if desired.
  Interventions: Other: Bio-mechanically correct manual therapy at the cervical atlanto-axial joints; Other: Bio-mechanically in-correct manual therapy at the cervical atlanto-axial joints
- Bio-mechanically incorrect manual therapy (received first) arm (Experimental): Participants will be randomized to receive manual therapy directed at the cervical spine atlanto-axial joints in the bio-mechanically incorrect direction followed by instruction in a home program to maintain this motion. Outcome measures will be assessed. Participants will return in 2-3 days and receive the opposite treatment and home program followed by outcomes assessment. Participants will return again in 2-3 days, outcomes will be assessed and the study will conclude. Participants will then be given the option to continue in formalized physical therapy if desired.
  Interventions: Other: Bio-mechanically correct manual therapy at the cervical atlanto-axial joints; Other: Bio-mechanically in-correct manual therapy at the cervical atlanto-axial joints

INTERVENTIONS:
Other: Bio-mechanically correct manual therapy at the cervical atlanto-axial joints — Participant is seated in a firm backed chair. The treating physical therapist mobilizes both the ipsi-lateral and contra-lateral atlanto-axial spinal segments congruently to the direction of rotational loss.
  Other Names: joint mobilization
Other: Bio-mechanically in-correct manual therapy at the cervical atlanto-axial joints — Participant is seated in a firm backed chair. The treating physical therapist mobilizes both the ipsi-lateral and contra-lateral atlanto-axial spinal segments in-congruently to the direction of rotational loss.
  Other Names: joint mobilization

SUMMARY:
Participants with limited neck rotation are recruited to determine if manual therapy (joint stretching) techniques applied in a bio-mechanically correct sequence will improve neck motion, function and pain better than if the manual therapy is applied in the opposite direction. Each participant will receive both the correct and the incorrect applications in randomized order with each treatment separated by 2-3 days. Improvement in neck motion, function and pain will be assessed after each session.

DETAILED DESCRIPTION:
Participants are recruited consecutively through referral from provider clinics or through self referral to physical therapy in the outpatient rehabilitation clinic at Indiana University Health West Hospital in Avon Indiana. After obtaining informed consent and meeting study criteria, participants will be randomized into either first receiving atlanto-axial joint mobilizations in a bio-mechanically correct or incorrect direction with respect to their loss of cervical rotation. Outcome measures will be completed both pre and post treatment. The participants will then be given self stretches at home to mimic the same intervention performed in the clinic three times per day. The participants will then return to the clinic in two or three days to receive the opposite treatment and opposite home program. Outcome data will again be collected both pre and post treatment. Participants will return for a final visit in two or three days and final outcome data will be collected and the participant will be offered continuation of physical therapy if neck symptoms still persist.

Planned Statistical Analysis:

* Descriptive statistics of subjects: age, gender, date of onset, Neck Disability Index, cervical active range of motion rotation, initial numeric pain rating at rest and rotating to the limited side
* Repeated measures ANOVA effect sizes for comparing differences between:

  1. Pre and post treatment comparing with-in treatment change for cervical range of motion rotation and numeric pain ratings on 1st and 2nd visits. Also comparing post treatment in cervical range of motion rotation and numeric pain ratings between 2nd and 3rd visits.
  2. Neck disability index change between 1st and 2nd visits and 2nd and 3rd visits
* Power calculation (actual achieved power)

ELIGIBILITY:
Inclusion Criteria:

* males or females between 18 and 80 years of age
* 25 percent or greater asymmetry of active cervical range of motion rotation limited by pain and/or stiffness

Exclusion Criteria:

* cervical surgeries or injections in the past one year
* current manual or exercise treatment by another provider for neck pain
* cervical manipulation/mobilization/trauma in past 3 months
* cervical radicular or referred pain distal to the acromion
* upper extremity neurologic myotome weakness or constant dermatomal numbness
* pending litigation
* signs of cervical myelopathy or vertebrobasilar artery insufficiency
* use of prescribed anticoagulants or documented blood clotting disorder
* alar or transverse ligament instability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
intra-visit change in cervical active range of motion rotation | day 1: pre and post treatment change, day 3: pre and post treatment change
  measured by standard goniometry

SECONDARY OUTCOMES:
intra-visit change in cervical pain at rest | day 1: pre and post treatment change, day 3: pre and post treatment change
  measured by the numeric pain rating scale 0-10
inter-visit change in neck disability/function | change between day 1 and day 3, change between day 3 and day 5
  measured by Neck Disability Index (NDI) score, range 0-100% with 0%= no disability and 100% = fully disabled
intra-visit change in cervical pain during most restricted active rotation | day 1: pre and post treatment change, day 3: pre and post treatment change
  measured by the numeric pain rating scale 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Michael Williams, MPT, Principal Investigator — Andrews University, Indiana University Health
Locations (1):
- Indiana University Health - West Hospital, Avon, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bishop MD, Mintken PE, Bialosky JE, Cleland JA. Patient expectations of benefit from interventions for neck pain and resulting influence on outcomes. J Orthop Sports Phys Ther. 2013;43(7):457-65. doi: 10.2519/jospt.2013.4492. Epub 2013 Mar 18. PMID 23508341
- [Background] Boyles R, Toy P, Mellon J Jr, Hayes M, Hammer B. Effectiveness of manual physical therapy in the treatment of cervical radiculopathy: a systematic review. J Man Manip Ther. 2011 Aug;19(3):135-42. doi: 10.1179/2042618611Y.0000000011. PMID 22851876
- [Background] Slaven EJ, Goode AP, Coronado RA, Poole C, Hegedus EJ. The relative effectiveness of segment specific level and non-specific level spinal joint mobilization on pain and range of motion: results of a systematic review and meta-analysis. J Man Manip Ther. 2013 Feb;21(1):7-17. doi: 10.1179/2042618612Y.0000000016. PMID 24421608
- [Background] Celenay ST, Akbayrak T, Kaya DO. A Comparison of the Effects of Stabilization Exercises Plus Manual Therapy to Those of Stabilization Exercises Alone in Patients With Nonspecific Mechanical Neck Pain: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2016 Feb;46(2):44-55. doi: 10.2519/jospt.2016.5979. Epub 2016 Jan 11. PMID 26755405
- [Background] van der Velde G, Yu H, Paulden M, Cote P, Varatharajan S, Shearer HM, Wong JJ, Randhawa K, Southerst D, Mior S, Sutton D, Jacobs C, Taylor-Vaisey A. Which interventions are cost-effective for the management of whiplash-associated and neck pain-associated disorders? A systematic review of the health economic literature by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Spine J. 2016 Dec;16(12):1582-1597. doi: 10.1016/j.spinee.2015.08.025. Epub 2015 Nov 26. PMID 26631759
- [Background] Schmid A, Brunner F, Wright A, Bachmann LM. Paradigm shift in manual therapy? Evidence for a central nervous system component in the response to passive cervical joint mobilisation. Man Ther. 2008 Oct;13(5):387-96. doi: 10.1016/j.math.2007.12.007. Epub 2008 Mar 3. PMID 18316238
- [Background] Creighton D, Gruca M, Marsh D, Murphy N. A comparison of two non-thrust mobilization techniques applied to the C7 segment in patients with restricted and painful cervical rotation. J Man Manip Ther. 2014 Nov;22(4):206-12. doi: 10.1179/2042618614Y.0000000077. PMID 25395829
- [Background] Aquino RL, Caires PM, Furtado FC, Loureiro AV, Ferreira PH, Ferreira ML. Applying Joint Mobilization at Different Cervical Vertebral Levels does not Influence Immediate Pain Reduction in Patients with Chronic Neck Pain: A Randomized Clinical Trial. J Man Manip Ther. 2009;17(2):95-100. doi: 10.1179/106698109790824686. PMID 20046551
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Background] Dunning JR, Cleland JA, Waldrop MA, Arnot CF, Young IA, Turner M, Sigurdsson G. Upper cervical and upper thoracic thrust manipulation versus nonthrust mobilization in patients with mechanical neck pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):5-18. doi: 10.2519/jospt.2012.3894. Epub 2011 Sep 30. PMID 21979312
- [Background] Youdas JW, Carey JR, Garrett TR. Reliability of measurements of cervical spine range of motion--comparison of three methods. Phys Ther. 1991 Feb;71(2):98-104; discussion 105-6. doi: 10.1093/ptj/71.2.98. PMID 1989013
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333